CLINICAL TRIAL: NCT04046510
Title: Comparaison of 3 Protocols of Ocytocin Administration in Cesarean Section
Brief Title: Comparaison of 3 Protocols of Ocytocin Administration in C Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor head of the anesthesia and intensive care department, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ocytocin in c section
Record Dates: First submitted 2019-07-31; First posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Cesarean Section Complications; Oxytocin Adverse Reaction
Keywords: Cesarean section, ocytocin, uterine tone, side effects
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: pre filled syringues of ocytocin were given to the care provider who didn't know the exact amount of ocytocin bolus and continious infusion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High doses (Active Comparator): the patients of this group recieved conventionnal doses of ocytocin after foetal extraction in C section: 5IU in bolus followed by 15IU in continuous infusion
  Interventions: Drug: Ocytocin
- Intermediate doses (Experimental): the patients of this group recieved after foetal extraction in C section: 2IU in bolus followed by 10IU in continuous infusion
  Interventions: Drug: Ocytocin
- Low doses (Experimental): the patients of this group recieved after foetal extraction in C section: 2IU in bolus followed by 5 IU in continuous infusion
  Interventions: Drug: Ocytocin

INTERVENTIONS:
Drug: Ocytocin — Administration of lower doses of Ocytocin in bolus and continuous infusion

SUMMARY:
This study aimed to compare 3 doses of ocytocin in bolus injection and contnious perfusion during C section. these doses determined by: high, intermediate and low doses, were administred to parturients during elective or urgent C section under spinal anesthesia

DETAILED DESCRIPTION:
This study aimed to compare 3 doses of ocytocin in bolus injection and contnious perfusion during C section. these doses determined by: high, intermediate and low doses, were administred to parturients during elective or urgent C section under spinal anesthesia.

The aim was to determine the lowest efficient dose to prevent post partum hemorrage and with the lowest incidence of maternal side effects.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients scheduled for C section under spinal anesthesia, monofoetal pregnancy, full term

Exclusion Criteria:

* necessity of general anesthesia
* non conscent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — including only parturients
Enrollment: 180 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
uterine tone | 10 minutes
  uterine tone juged by the obstetrician

SECONDARY OUTCOMES:
hemoglobin rate | 30 minutes after C section
  delta hemoglobin: preoperative HB- Post operative HB
Additive boluses of Ocytocin | 30 minutes after C section
  necessity of Additive boluses of Ocytocin
side effects of Ocytocin | up to 30 minutes after C section
  Tachycardia, hypotension, nausea vomiting, headache, chest pain

CONTACTS AND LOCATIONS:
Locations (1):
- Mongi Slim Hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided